CLINICAL TRIAL: NCT02472132
Title: The Use of Point of Care Ultra Sound for Correct Placement of Central Venous Catheter and for the Detection of Complications
Brief Title: The Use of Point of Care Ultra Sound for Correct Placement of Central Venous Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SOR-0131-15-CTIL
Record Dates: First submitted 2015-05-18; First posted 2015-06-15 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Central Venous Catheter
Keywords: Central Venous Catheter; Point Of Care Ultra Sound; Sub Clavian Vein; Internal Jugular Vein; Trans Thoracic Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Prospective implantation of POC US for CVC tip placement.
  Interventions: Device: POC US
- Control (No Intervention): Retrospective data collection for CVC placement in the medical and surgical ICUs, before the initiation of the study and without the use of POCUS for CVC tip placement.

INTERVENTIONS:
Device: POC US — Use of point of care ultrasound in insertion of CVC
  Arms: Intervention

SUMMARY:
Central venous catheter (CVC) is an essential tool in the management of both medical and surgical patients. Establishing venous access is critically important and is sometimes technically challenging. Among the many indications for point of care ultrasound (POCUS), ultrasound-guided venous catheter placement is well described and increasingly used. This study was designed to evaluate the utility of peri procedural transthoracic echocardiography (TTE) as a tool for positioning CVC and for ruling out complications.

DETAILED DESCRIPTION:
Central venous catheter (CVC) is an essential tool in the management of both medical and surgical patients. Establishing venous access is critically important and is sometimes technically challenging. Among the many indications for point of care ultrasound (POCUS), ultrasound-guided venous catheter placement is well described and increasingly used. This study was designed to evaluate the utility of peri procedural transthoracic echocardiography (TTE) as a tool for positioning CVC and for ruling out complications.

The study population will be screened at the internal wards and medical intensive care unit of Soroka Medical Center.

Research candidates' files will be screened routinely by a study coordinator. The study population will be enrolled according to the inclusion and exclusion criteria.

The primary objective for the study is to evaluate whether the use of POCUS in CVC insertion can help inaccurate CVC tip placement, detect misplacement and complications and better than chest X ray.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to internal ward or medical intensive care unit
2. Patients in need for central venous catheter in the subclavian or internal jugular veins

Exclusion Criteria:

1. Subject currently enrolled in another investigational study
2. Surgical patients with open abdomen covered with bogota bag or vac - pac
3. Patients with pneumothorax prior to central venous catheter insertion
4. Patients in need for central venous catheter for hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Rate of misplacement of the tip of CVC. | 6 months

SECONDARY OUTCOMES:
Rate of ventricular arrhythmia during line insertion while using POC US | 6 months
Duration time of CVC insertion using POC US | 6 months
Number of CVC insertion complications using POC US | 6 months
Sensitivity (score-the device's ability to identify a condition correctly) of POC US in detection of CVC insertion complications | 6 months
Specificity (score-the device's ability to exclude a condition correctly) of POC US in detection of CVC insertion complications | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Byon HJ, Lee GW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Comparison between ultrasound-guided supraclavicular and infraclavicular approaches for subclavian venous catheterization in children--a randomized trial. Br J Anaesth. 2013 Nov;111(5):788-92. doi: 10.1093/bja/aet202. Epub 2013 Jun 10. PMID 23756247
- [Result] Troianos CA, Hartman GS, Glas KE, Skubas NJ, Eberhardt RT, Walker JD, Reeves ST; Councils on Intraoperative Echocardiography and Vascular Ultrasound of the American Society of Echocardiography; Society of Cardiovascular Anesthesiologists. Special articles: guidelines for performing ultrasound guided vascular cannulation: recommendations of the American Society of Echocardiography and the Society Of Cardiovascular Anesthesiologists. Anesth Analg. 2012 Jan;114(1):46-72. doi: 10.1213/ANE.0b013e3182407cd8. Epub 2011 Nov 29. No abstract available. PMID 22127816
- [Result] Levy JA, Noble VE. Bedside ultrasound in pediatric emergency medicine. Pediatrics. 2008 May;121(5):e1404-12. doi: 10.1542/peds.2007-1816. PMID 18450883
- [Result] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Result] Rabindranath KS, Kumar E, Shail R, Vaux E. Use of real-time ultrasound guidance for the placement of hemodialysis catheters: a systematic review and meta-analysis of randomized controlled trials. Am J Kidney Dis. 2011 Dec;58(6):964-70. doi: 10.1053/j.ajkd.2011.07.025. PMID 22099570
- [Result] Sigaut S, Skhiri A, Stany I, Golmar J, Nivoche Y, Constant I, Murat I, Dahmani S. Ultrasound guided internal jugular vein access in children and infant: a meta-analysis of published studies. Paediatr Anaesth. 2009 Dec;19(12):1199-206. doi: 10.1111/j.1460-9592.2009.03171.x. Epub 2009 Oct 23. PMID 19863734
- [Result] Bedel J, Vallee F, Mari A, Riu B, Planquette B, Geeraerts T, Genestal M, Minville V, Fourcade O. Guidewire localization by transthoracic echocardiography during central venous catheter insertion: a periprocedural method to evaluate catheter placement. Intensive Care Med. 2013 Nov;39(11):1932-7. doi: 10.1007/s00134-013-3097-3. Epub 2013 Sep 20. PMID 24052186
- [Result] Gillman LM, Blaivas M, Lord J, Al-Kadi A, Kirkpatrick AW. Ultrasound confirmation of guidewire position may eliminate accidental arterial dilatation during central venous cannulation. Scand J Trauma Resusc Emerg Med. 2010 Jul 13;18:39. doi: 10.1186/1757-7241-18-39. PMID 20626896
- [Result] Hocking G. Central venous access and monitoring. Practical Procedures 2000;12:1-6.
- [Result] Sznajder JI, Zveibil FR, Bitterman H, Weiner P, Bursztein S. Central vein catheterization. Failure and complication rates by three percutaneous approaches. Arch Intern Med. 1986 Feb;146(2):259-61. doi: 10.1001/archinte.146.2.259. PMID 3947185
- [Result] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399
- [Result] Prekker ME, Chang R, Cole JB, Reardon R. Rapid confirmation of central venous catheter placement using an ultrasonographic "Bubble Test". Acad Emerg Med. 2010 Jul;17(7):e85-6. doi: 10.1111/j.1553-2712.2010.00785.x. No abstract available. PMID 20653578
- [Result] Vezzani A, Brusasco C, Palermo S, Launo C, Mergoni M, Corradi F. Ultrasound localization of central vein catheter and detection of postprocedural pneumothorax: an alternative to chest radiography. Crit Care Med. 2010 Feb;38(2):533-8. doi: 10.1097/CCM.0b013e3181c0328f. PMID 19829102
- [Result] Merrer J, De Jonghe B, Golliot F, Lefrant JY, Raffy B, Barre E, Rigaud JP, Casciani D, Misset B, Bosquet C, Outin H, Brun-Buisson C, Nitenberg G; French Catheter Study Group in Intensive Care. Complications of femoral and subclavian venous catheterization in critically ill patients: a randomized controlled trial. JAMA. 2001 Aug 8;286(6):700-7. doi: 10.1001/jama.286.6.700. PMID 11495620
- [Result] Ullman JI, Stoelting RK. Internal jugular vein location with the ultrasound Doppler blood flow detector. Anesth Analg. 1978 Jan-Feb;57(1):118. doi: 10.1213/00000539-197801000-00024. No abstract available. PMID 564628
- [Result] Lichtenstein DA, Menu Y. A bedside ultrasound sign ruling out pneumothorax in the critically ill. Lung sliding. Chest. 1995 Nov;108(5):1345-8. doi: 10.1378/chest.108.5.1345. PMID 7587439
- [Result] Lichtenstein D, Meziere G, Biderman P, Gepner A. The comet-tail artifact: an ultrasound sign ruling out pneumothorax. Intensive Care Med. 1999 Apr;25(4):383-8. doi: 10.1007/s001340050862. PMID 10342512
- [Result] Maury E, Guglielminotti J, Alzieu M, Guidet B, Offenstadt G. Ultrasonic examination: an alternative to chest radiography after central venous catheter insertion? Am J Respir Crit Care Med. 2001 Aug 1;164(3):403-5. doi: 10.1164/ajrccm.164.3.2009042. PMID 11500340